CLINICAL TRIAL: NCT07354815
Title: Determination of the Level of Correlation Between Periodontal Inflammatory Surface Area and Metabolic Syndrome-Associated Periodontal Tissue Destruction
Brief Title: Metabolic Syndrome-Associated Periodontal Inflammatory Surface Area
Status: Not yet recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek KARADOĞAN, Assoc. Prof. Dr., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: MetSPISA07/2025
Record Dates: First submitted 2025-08-28; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Syndrome (MetS); Periodontitis
Keywords: metabolic syndrome; periodontitis; periodontal inflammatory surface area
MeSH Terms: conditions — Metabolic Syndrome; Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Serum blood samples Routine blood tests will include fasting blood glucose, HbA1c, triglyceride, HDL, and hsCRP levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with metabolic syndrome: Metabolic syndrome is diagnosed according to the National Cholesterol Education Program Adult Treatment Panel III (NCEP/ATP III) criteria. Diagnosis is made by meeting three of the following five criteria: waist circumference: ≥ 94 cm in men and ≥ 88 cm in women, blood pressure ≥ 130/85 mmHg or use of antihypertensive medication, fasting blood glucose ≥ 100 mg/dL or diagnosed type 2 diabetes, triglycerides ≥ 1.7 mmol/L, and HDL < 1.29 mmol/L.

SUMMARY:
This study aims to examine the potential of metabolic syndrome (MetS), a systemic, inflammatory disease, to influence the relationship between periodontal inflammatory surface area (PISA) and diabetes and obesity parameters. The primary question addressed by the study is:

Can PISA be used as a significant parameter in the relationship between periodontal disease and MetS? In this context, the relationship between PISA and periodontal clinical parameters and serum parameters directly related to the diagnosis of MetS will be examined.

DETAILED DESCRIPTION:
This study aims to investigate the potential of metabolic syndrome (MetS), a systemic and inflammatory disease, to influence the relationship between periodontal inflammatory surface area (PISA) and diabetes and obesity parameters. Our hypothesis will test whether PISA can be used as a significant parameter in the relationship between periodontal disease and MetS. This cross-sectional study will examine the relationship between PISA and other periodontal clinical parameters (plaque index (PI), bleeding on probing (BPO), probing pocket depth (SCD), clinical attachment loss (CAL)), serum HbA1c, fasting blood glucose, lipid profile (HDL and triglyceride levels), body mass index (BMI), and hsCRP, which are directly related to MetS diagnosis, in patients with MetS.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years of age
* Presence of at least three of the following parameters: (For MetS diagnosis) Waist circumference: ≥ 94 cm for men, ≥ 88 cm for women Blood pressure ≥ 130/85 mmHg or taking antihypertensive medication Fasting blood glucose ≥ 100 mg/dl or diagnosed with Type 2 Diabetes Triglycerides ≥ 1.7 mmol/L HDL < 1.29 mmol/L
* Having at least 20 teeth
* Not having received periodontal therapy in the last 6 months
* Not having taken antibiotics, steroids, and/or nonsteroidal anti-inflammatory drugs in the last 3 weeks
* Not having any autoimmune disease, osteoporosis, or cancer
* Not taking immunosuppressive medications, oral contraceptives, Not taking bisphosphonates
* Not being pregnant
* Not having an active infectious disease (acute hepatitis, tuberculosis, AIDS)
* Not taking chronic medications that affect periodontal tissues (cyclosporine A, phenytoin)
* Not taking antioxidant supplements in the last 6 months

Exclusion Criteria:

* Patients with active infectious disease,
* Those taking medications that may affect periodontal tissues,
* Those who did not sign the informed consent form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metabolic syndrome who come to the Periodontology Clinic of Recep Tayyip Erdoğan University Faculty of Dentistry for routine periodontal treatment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Periodontal Inflammatory Surface Area (PISA) Calculation | Day 1
  PISA is automatically obtained by transferring the bleeding on probing (BOP), clinical attachment loss (CAL) and gingival recession measured from 6 regions (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) of each tooth into a Microsoft Excel spreadsheet.
  Bleeding on Probing (BOP):
  Bleeding from the gingival tissue occurs as a result of light force applied to the periodontal pocket during probing. It is often an early indicator of gingival inflammation and is used to determine periodontal disease activity.
  Clinical Attachment Loss (CAL):
  This is the distance from the gingival margin to the cemento-cemental junction, measured with a periodontal probe. It refers to the loss of periodontal supporting tissues (periodontal ligament and alveolar bone) and is used to assess the severity of periodontal disease.
  Gingival Recession:
  This is the displacement of the gingival margin apically toward the cemento-cemental junction.

SECONDARY OUTCOMES:
Clinical Periodontal Parameters (Plaque Index) | Day 1
  Plaque Index (PI) (Silness and Löe, 1964) This index is used to evaluate the amount of dental plaque accumulation on tooth surfaces. Each tooth's four surfaces (buccal, lingual, mesial, distal) are examined using a probe or visually. Each surface is scored from 0 to 3. The average score is calculated for each tooth. The overall plaque index is obtained by averaging the scores from all examined teeth.
  Score Description 0 No plaque.
  1. No visible plaque, but a slight film of plaque is detected when a probe is run along the gingival margin.
  2. Visible plaque along the gingival margin, forming a continuous band.
  3. Abundant plaque covering the gingival area and extending toward the middle of the tooth surface, including the interproximal spaces.
Periodontal Clinical Parametres (Bleeding on Probing Index) | Day 1
  This index is used to assess the presence and severity of gingival inflammation by observing bleeding after gentle pressure is applied to the gingival sulcus using a periodontal probe. A thin periodontal probe is gently inserted into the gingival sulcus with light pressure (approximately 20-25 grams). Bleeding occurring within 10-30 seconds is observed. Each measurement site is recorded as either "bleeding present" or "bleeding absent." Presence of bleeding is an early and sensitive indicator of gingival inflammation.
  Score Description:
  0 No bleeding
  1 Bleeding present (mild or severe)
Periodontal Clinical Parametres (Probing Pocket Depth) | Day 1
  Using a Williams periodontal probe, the distance between the gingival margin and the base of the periodontal pocket is measured in millimeters at six sites per tooth: mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual. All teeth are measured. The values obtained from each site are summed and then divided by the total number of sites measured. This gives the average probing depth for the individual.
  Measurement Interpretation 1-3 mm Healthy sulcus 4-5 mm Shallow to moderate pocket
  ≥6 mm Deep periodontal pocket (advanced disease)
Periodontal Clinical Parametres (Clinical Attachment Loss) | Day 1
  Using a Williams periodontal probe, the distance between the enamel-cementum junction and the base of the periodontal pocket is measured in millimeters at six sites per tooth: mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual. All teeth are measured. The values obtained from each site are summed and then divided by the total number of sites measured. This gives the average probing depth for the individual.
  CAL Value Interpretation 0-1 mm Healthy / minimal loss 2-3 mm Mild attachment loss 4-5 mm Moderate attachment loss
  ≥6 mm Severe attachment loss
Sociodemographic Data | Day 1
  Sociodemographic data, including patients' age, gender, smoking, socioeconomic status, education level, and how many times a day they brush their teeth, will be noted.

OTHER OUTCOMES:
Fasting blood glucose | Day 1
  Fasting Blood Glucose: The plasma glucose concentration measured after at least 8 hours of caloric restriction. It is a fundamental biochemical parameter for assessing glycemic status and diagnosing diabetes.
Glycated Hemoglobin A1c | Day 1
  HbA1c (Glycated Hemoglobin A1c): A stable complex formed by the non-enzymatic covalent binding of glucose to the β-chain of hemoglobin, reflecting the average blood glucose level over the lifespan of erythrocytes (approximately 120 days). It is considered a gold standard indicator of long-term glycemic control.
Triglyceride | Day 1
  Triglyceride: A neutral lipid composed of three fatty acids esterified to a glycerol backbone. It is primarily transported in plasma by VLDL and chylomicrons and serves as a biomarker of dyslipidemia and cardiometabolic risk.
HDL (High-Density Lipoprotein) | Day 1
  HDL (High-Density Lipoprotein): Lipoprotein particles of high density that play a central role in reverse cholesterol transport, shuttling cholesterol from peripheral tissues to the liver for excretion. They exhibit anti-atherogenic, anti-inflammatory, and antioxidant properties.
hsCRP (High-Sensitivity C-Reactive Protein) | Day 1
  hsCRP (High-Sensitivity C-Reactive Protein): The low-level concentrations of the liver-derived acute-phase reactant CRP, measured by high-sensitivity immunoturbidimetric or nephelometric assays. It serves as a biomarker of subclinical inflammation and cardiovascular risk.
Waist Circumference | Day 1
  Waist Circumference: The individual stands upright. A tape measure is taken horizontally at the narrowest point of the waist (usually between the bottom of the ribs and the top of the hipbone).
Height | Day 1
  Height: a measure of vertical distance, vertical dimension, or vertical position.
Weight | Day 1
  Weight is the gravitational force exerted on an object.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology of the Faculty of Dentistry of Recep Tayyip Erdogan University, Rize, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No